CLINICAL TRIAL: NCT04048057
Title: The Effect of Different Exercise Programs in Coronary Artery Patients: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Okur, Kutahya Medical Sciences University, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMSU-Exercise
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Exercise; Cardiac Rehabilitation
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modarete Intensity Continous Training (Experimental)
  Interventions: Other: Exercise
- High Intensity Interval Training I (Experimental)
  Interventions: Other: Exercise
- High Intensity Interval Training II (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Modarete Intensity Continous Training: Medium intensity continuous exercise training will be performed. Exercise intensity will be adjusted as 50-70% of maximal power.
  High Intensity Interval Training I: It will be four cycles consisting of 4 minute high intensity exercise phase and 3 minute active recovery phase. High intensity phase will be adjusted as 85-100% of maximal power and active recovery phase as 50-70% of maximal power.
  High Intensity Interval Training II: It will be 10 cycles consisting of 1 minute high intensity exercise phase and 1 minute active recovery phase. High intensity phase will be adjusted as 85-100% of maximal power and active recovery phase as 50-70% of maximal power.

SUMMARY:
There are studies showing the superiority of HIIT protocols in patients with CAD in the literature, however there is no consensus on the use of HIIT protocols in CAD patients. In addition, in these studies, the HIIT protocols differ in severity and duration and there is no optimal HIIT protocol. Therefore, this study was planed to investigate of two different HIIT protocols and one MICT protocols, which are more commonly used in patients with CAD in the literature on exercise capacity, quality of life, body composition, physical activity level and fear of movement.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone percutaneous transluminal coronary angioplasty or coronary artery bypass graft surgery,
* Nonobstructive CAD registered by angiography
* Left ventricular ejection fraction above 50%,
* Clinically stable for more than 2 weeks in terms of symptoms and medical treatment.

Exclusion Criteria:

* Ischemia symptoms,
* Being in Class III-IV according to the New York Heart Classification,
* Obtaining significant left ventricular outflow obstruction,
* Ventricular arrhythmia,
* Being marked valvular heart disease,
* Failure to comply with exercise testing and training rules,
* To have significant orthopedic or neurological comorbidity that prevents full participation.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
exercise capacity | 15 minutes
  Cardiopulmonary exercise test

SECONDARY OUTCOMES:
MacNew Health Related Quallity of Life Qustionnaire | 15 minutes
  The validity and reliability of the MacNew Heart Disease Health-Related Quality of Life Questionnaire Daşkapan et al. in 2008. It is a scale developed to determine the quality of life in heart diseases consisting of 27 items each containing a 7-point Likert type response. In the evaluation of the scale, 3 sub-dimensions (emotional, physical and social) and total score values are used
body composition | 1 minute
  Tanita
physical activity level | 15 minutes
  International Physical Activity Questionnaire
fear of movement | 15 minutes
  Tampa

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided